CLINICAL TRIAL: NCT03231735
Title: A Randomized Controlled Trial of Mid and Standard Frequency Ventilation in Infants With Respiratory Distress Syndrome
Brief Title: Mid and Standard Frequency Ventilation in Infants With Respiratory Distress Syndrome
Acronym: MIDAS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of South Alabama (Other)
Responsible Party: Principal Investigator, Colm Travers, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F160701002
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Ventilator-Induced Lung Injury; Respiratory Distress Syndrome; Bronchopulmonary Dysplasia; Preterm Infant
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Respiratory Distress Syndrome; Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial with a 1:1 parallel allocation of infants to mid or standard frequency ventilation using stratified permuted block design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mid frequency ventilation (Other): Mid frequency ventilation delivered at rates > 60 per minute and ≤ 150 per minute, with patient triggered ventilation and pressure support.
  Interventions: Device: Mid frequency ventilation
- Standard frequency ventilation (Other): Standard frequency ventilation delivered at rates < 60 per minute and ≥ 20 per minute, with patient triggered ventilation and pressure support.
  Interventions: Device: Standard frequency ventilation

INTERVENTIONS:
Device: Mid frequency ventilation — Mechanical ventilator used at rates > 60 per minute and ≤ 150 per minute, with patient triggered ventilation and pressure support.
  Arms: Mid frequency ventilation
Device: Standard frequency ventilation — Mechanical ventilator used at rates < 60 per minute and ≥ 20 per minute, with patient triggered ventilation and pressure support.
  Arms: Standard frequency ventilation

SUMMARY:
The purpose of this study is to determine, in preterm infants less than 37 weeks gestation with respiratory distress who are ventilated in the first 48 hours after birth, if mid frequency ventilation strategy using ventilator rate of ≥ 60 to ≤ 150 per minute compared with standard frequency ventilation strategy using ventilator rates of ≥ 20 to < 60 per minute will increase the number of alive ventilator-free days after randomization and reduce the risk of ventilator induced lung injury.

DETAILED DESCRIPTION:
In preterm infants with respiratory distress syndrome (RDS) who are ventilated in the first 48 hours after birth, mid frequency ventilation (MFV) strategy, compared with standard frequency ventilation (SFV) strategy, in the first week after birth, will increase the number of days alive and ventilator-free in the 28 days after birth.

This will be a randomized controlled trial with a 1:1 parallel allocation of infants to MFV or SFV using stratified permuted block design. Randomization will be stratified by gestational age (≥ 23 weeks to ˂ 26 weeks, ≥ 26 weeks to ≤ 28+6/7 (less than 29 weeks), and 29+0/7 to 36+6/7). Randomization of twins and higher orders (when eligible) will be to the same group.

Inborn and outborn infants who are receiving assisted ventilation for RDS in the first 48 hours after birth will be included in this study. Infants with any of the following: a major malformation, a neuromuscular condition that affects respiration, terminal illness or decision to withhold or limit support will not be eligible.

Infants will be randomized to MFV versus SFV. MFV delivered at rates > 60 per minute and ≤ 150 per minute, with patient triggered ventilation and pressure support.

SFV delivered at rates < 60 per minute and ≥ 20 per minute, with patient triggered ventilation and pressure support.

ELIGIBILITY:
Inclusion Criteria:

* Infants ≥ 23+0/7 weeks and ≤ 36+6/7 who are intubated and mechanically ventilated for respiratory distress syndrome (defined by use of surfactant) within 48 hours after birth
* Infants whose parents/legal guardians have provided consent for enrollment
* Inborn or outborn infants transferred to this center before 48 hours after birth
* Ventilator rate ≤ 80 per minute prior to enrollment

Exclusion Criteria:

* a major malformation, a neuromuscular condition that affects respiration, or terminal illness or decision to withhold or limit support.

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2021-11-21 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Alive ventilator free days | Days 1-28 after birth
  The number of days alive and ventilator-free

SECONDARY OUTCOMES:
Alive at day 28 after birth | Day 28 after birth
  Number of infants alive
Ventilator free | Day 28 after birth
  Number of infants ventilator free
Bronchopulmonary dysplasia | Measured at 36 weeks' postmenstrual age
  Bronchopulmonary dysplasia in preterm infants less than 32 weeks' gestation
Bronchopulmonary dysplasia | Measured at 36 weeks' postmenstrual age
  Bronchopulmonary dysplasia in preterm infants less than 29 weeks' gestation
Air leak syndrome | Day 1-28 after birth
  Rate of pulmonary interstitial emphysema and/or pneumothorax
Pulmonary hemorrhage | Day 1-28 after birth
  Rate of pulmonary hemorrhage
Severe (grade 3-4) intracranial hemorrhage | Day 1-30 after birth
  Rate of severe (grade 3-4) intracranial hemorrhage in infants less than 29 weeks' gestation
Alive and continuous positive airway pressure/ventilator free | Day 1-28 after birth
  Number of days alive and ontinuous positive airway pressure/ventilator free
Alive and oxygen free | Day 1-28 after birth
  Number of days alive and oxygen free
Postnatal steroids | Before 36 weeks' postmenstrual age
  Rate of post natal steroids for bronchopulmonary dysplasia
Necrotizing enterocolitis | Days 1-120 after birth
  Rate of proven necrotizing enterocolitis (NEC) in infants less than 29 weeks' gestation
Neurodevelopmental impairment | 18 to 24 months after birth
  Rate of moderate to severe neurodevelopmental impairment in survivors < 27 weeks' gestation
Bronchopulmonary dysplasia or death | Day 1-120 after birth
  Rate of Bronchopulmonary dysplasia or death
Neurodevelopmental impairment or death | Day 1-120 after birth
  Rate of Bronchopulmonary dysplasia or death
Bronchopulmonary dysplasia or death | 18 to 24 months after birth
  Rate of moderate to severe neurodevelopmental impairment or death
Necrotizing enterocolitis or death | Day 1-120 after birth
  Rate of proven necrotizing enterocolitis or death
Death | Day 1-120 after birth
  Death before hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar A Carlo, MD, Study Director — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama, Mobile, Alabama

IPD SHARING:
Plan to Share IPD: No